CLINICAL TRIAL: NCT06989671
Title: A Phase 2 Study of SYS6002 in Combination With JMT101 and Enlonstobart Injection in Participants With Recurrent and/or Metastatic Head and Neck Squamous Cell Cancer (HNSCC)
Brief Title: SYS6002 Plus JMT101 and Enlonstobart Injection in Participants With HNSCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC Megalith Biopharmaceutical Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SYS6002-003
Record Dates: First submitted 2025-04-25; First posted 2025-05-25 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, factorial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- SYS6002 monotherapy (Q2W) (Experimental)
  Interventions: Drug: SYS6002
- SYS6002 monotherapy (Q3W) (Experimental)
  Interventions: Drug: SYS6002
- JMT101 monotherapy (Experimental)
  Interventions: Drug: JMT101
- SYS6002 combinational therapy (Q2W) (Experimental)
  Interventions: Drug: JMT101; Drug: SYS6002; Drug: SG001
- SYS6002 combinational therapy (Q3W) (Experimental)
  Interventions: Drug: JMT101; Drug: SYS6002; Drug: SG001
- Factorial Group (Experimental)
  Interventions: Drug: SYS6002; Drug: SG001
- Experimental Group 1 (Experimental)
  Interventions: Drug: JMT101; Drug: SYS6002; Drug: SG001
- Experimental Group 2 (Experimental)
  Interventions: Drug: JMT101; Drug: SYS6002; Drug: SG001

INTERVENTIONS:
Drug: JMT101 — JMT101 Q2W or Q3W, intravenous injection
  Arms: Experimental Group 1; Experimental Group 2; JMT101 monotherapy; SYS6002 combinational therapy (Q2W); SYS6002 combinational therapy (Q3W)
Drug: SYS6002 — SYS6002 Q2W or Q3W, intravenous injection
  Arms: Experimental Group 1; Experimental Group 2; Factorial Group; SYS6002 combinational therapy (Q2W); SYS6002 combinational therapy (Q3W); SYS6002 monotherapy (Q2W); SYS6002 monotherapy (Q3W)
Drug: SG001 — SG001 Q2W or Q3W, intravenous injection
  Arms: Experimental Group 1; Experimental Group 2; Factorial Group; SYS6002 combinational therapy (Q2W); SYS6002 combinational therapy (Q3W)

SUMMARY:
This is a Phase II study of anti-nectin-4 ADC combined with the EGFR monoclonal antibody and the PD-1 monoclonal antibody in participants with advanced head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
This trial consists of two parts. Part 1 (Monotherapy Group) evaluates both SYS6002 monotherapy (stratified into two cohorts by dose levels and administration frequencies) and JMT101 monotherapy. Part 2 (Combination Therapy Group) comprises Stage 1 (dose escalation phase) and Stage 2 (proof-of-concept phase). Following completion of the dose escalation phase in Part 2 and evaluation of integrated efficacy and safety analyses of SYS6002 monotherapy in Part 1 of this study as well as other clinical studies involving participants with ≥2L HNSCC, the decision on progressing to Stage 2 of Part 2 will be made through discussion between the Sponsor and investigators.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older, regardless of gender.
* Able to understand and voluntarily sign a written informed consent form (ICF).
* Confirmed recurrent or metastatic HNSCC that is not curable with local treatments. Primary tumor must be located in the oral cavity, oropharynx, hypopharynx, or larynx.
* Able to provide well-preserved or fresh tumor tissue.
* According to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, at least one measurable lesion confirmed by CT or MRI.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1.
* Life expectancy ≥ 3 months.
* Normal major organ function within 7 days prior to treatment.

Exclusion Criteria:

* Primary tumor located in the nasopharynx, nasal cavity, paranasal sinuses, salivary glands, thyroid or parathyroid glands, skin, or squamous cell carcinoma with an unknown primary site.
* Presence of leptomeningeal metastasis, spinal cord compression, symptomatic or progressive brain metastases.
* (Only for Stage 2 in Part 2) Prior systemic anti-tumor therapy for recurrent or metastatic HNSCC.
* Known allergy to any component of SYS6002, JMT101, or Enlonstobart injection.
* Participants who have previously received MMAE toxin ADC treatment (only for Part 1 and Stage 2 in Part 2).
* Adverse events related to prior anti-tumor treatment that have not resolved to ≤ Grade 1 according to NCI-CTCAE v5.0 (except for toxicities deemed low-risk by the investigator, such as Grade 2 alopecia).
* Washout period not met for anti-tumor medications or treatments.
* Any serious and/or uncontrolled comorbid conditions that may interfere with the participant's ability to participate in the study
* Pregnant or breastfeeding women; women of childbearing potential with a positive pregnancy test within 7 days before enrollment. Breastfeeding women may participate if they stop breastfeeding, but they cannot resume breastfeeding during the treatment and after the study ends.
* Any male or female participants of childbearing potential who refuse to use highly effective contraception during the study and for 6 months after the last dose of study drug.
* Unwilling or unable to comply with the study procedures and requirements, or deemed unsuitable for participation by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicities (DLTs) | Up to 28 days
Incidence of Adverse Events (AEs) | Up to approximately 2 years
Maximum Tolerated Dose (MTD) | Up to approximately 2 years
Objective Response Rate (ORR) | Up to approximately 2 years

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to approximately 2 years
Duration of Response (DOR) | Up to approximately 2 years
Progression-free Survival (PFS) | Up to approximately 2 years
Overall Survival (OS) | Up to approximately 3 years